CLINICAL TRIAL: NCT03038399
Title: A 24-month Phase II Open-label, Multicenter Long-term Extension Study to Assess the Long-Term Safety and Efficacy of Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: Long-term Extension Study to Assess Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Collaborators: University of Pittsburgh (Other); Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VBP15-LTE
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; vamorolone
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level Group 1 (Experimental): Participants enrolled in Dose Level Group 1 will receive vamorolone 0.25 mg/kg/day.
  Interventions: Drug: Vamorolone 0.25 mg/day/day
- Dose Level Group 2 (Experimental): Participants enrolled in Dose Level Group 2 will receive vamorolone 0.75 mg/kg/day.
  Interventions: Drug: Vamorolone 0.75 mg/day/day
- Dose Level Group 3 (Experimental): Participants enrolled in Dose Level Group 3 will receive vamorolone 2.0 mg/kg/day.
  Interventions: Drug: Vamorolone 2.0 mg/day/day
- Dose Level Group 4 (Experimental): Participants enrolled in Dose Level Group 4 will receive vamorolone 6.0 mg/kg/day.
  Interventions: Drug: Vamorolone 6.0 mg/day/day

INTERVENTIONS:
Drug: Vamorolone 0.25 mg/day/day — Oral administration of 0.25 mg/kg/day daily for 24 months.
  Other Names: VBP15
  Arms: Dose Level Group 1
Drug: Vamorolone 0.75 mg/day/day — Oral administration of 0.75 mg/kg/day daily for 24 months.
  Other Names: VBP15
  Arms: Dose Level Group 2
Drug: Vamorolone 2.0 mg/day/day — Oral administration of 2.0 mg/kg/day daily for 24 months.
  Other Names: VBP15
  Arms: Dose Level Group 3
Drug: Vamorolone 6.0 mg/day/day — Oral administration of 6.0 mg/kg/day daily for 24 months.
  Other Names: VBP15
  Arms: Dose Level Group 4

SUMMARY:
This long-term extension study is an open-label, multiple-dose study to evaluate the long-term safety, tolerability, efficacy and PD of vamorolone administered once daily by liquid oral suspension over a Treatment Period of 24 months to young boys with DMD who participated in the VBP15-002 Phase IIa and VBP15-003 Phase IIa extension core studies.

DETAILED DESCRIPTION:
This study will evaluate if it is safe to use a new medication called vamorolone for more than two weeks in children with DMD, if boys with DMD who take the study medication have improved muscle function compared to boys with DMD in other studies who did not take any type of steroid, and to see if boys with DMD who take the study medication gain less weight compared to boys with DMD in a prior study who took another type of steroid called prednisone. Enrolled participants will take the study medication for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent or legal guardian has provided written informed consent and HIPAA authorization (if applicable) prior to any VBP15-LTE long-term extension study-specific procedures;
2. Subject has previously completed study VBP15-003 up to and including the Week 24 Final assessments, prior to enrolling in the VBP15-LTE study at the conclusion of the VBP15-003 Week 24 Visit [Note: if entering the dose-tapering period, subject is enrolling within 8 weeks after the VBP15-003 final visit following dose-tapering]; and
3. Subject and parent/guardian are willing and able to comply with scheduled visits, study drug administration plan, and study procedures.

Exclusion Criteria:

1. Subject had a serious or severe adverse event in study VBP15-003 that, in the opinion of the Investigator, was probably or definitely related to vamorolone use and precludes safe use of vamorolone for the subject in this long-term extension study;
2. Subject has current or history of major renal or hepatic impairment, diabetes mellitus or immunosuppression;
3. Subject has current or history of chronic systemic fungal or viral infections;
4. Subject has used mineralocorticoid receptor agents, such as spironolactone, eplerenone, canrenone (canrenoate potassium), prorenone (prorenoate potassium), mexrenone (mexrenoate potassium) within 4 weeks prior to the first dose of study medication;
5. Subject has evidence of symptomatic cardiomyopathy. [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
6. Subject is currently being treated or has received previous treatment with oral glucocorticoids or other immunosuppressive agents [Notes: Past transient use of oral glucocorticoids or other oral immunosuppressive agents for no longer than 3 months cumulative, with last use at least 3 months prior to first dose of study medication, will be considered for eligibility on a case-by-case basis. Inhaled and/or topical glucocorticoids prescribed for an indication other than DMD are permitted but must be administered at stable dose for at least 3 months prior to study drug administration];
7. Subject has used idebenone within 4 weeks prior to the first dose of study medication;
8. Subject has an allergy or hypersensitivity to the study medication or to any of its constituents;
9. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
10. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator
11. Subject is currently taking any investigational drug, or has taken any investigational drug other than vamorolone within 3 months prior to the start of study treatment.

Note: Subjects may be re-evaluated if ineligible due to a transient condition which would prevent the subject from participating.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Clemens, MD, Study Chair — University of Pittsburgh
Locations (12):
- United States (6):
  - University of California Davis, Davis, California
  - University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - Royal Children's Hospital, Melbourne
  - Sydney Children's Hospital, Westmead
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Schneider Children's Medical Center, Petah Tikva, Israel
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Smith EC, Conklin LS, Hoffman EP, Clemens PR, Mah JK, Finkel RS, Guglieri M, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, Kerchner L, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, Gordish-Dressman H, Hagerty L, Dang UJ, Damsker JM, Schwartz BD, Mengle-Gaw LJ, McDonald CM; CINRG VBP15 and DNHS Investigators. Efficacy and safety of vamorolone in Duchenne muscular dystrophy: An 18-month interim analysis of a non-randomized open-label extension study. PLoS Med. 2020 Sep 21;17(9):e1003222. doi: 10.1371/journal.pmed.1003222. eCollection 2020 Sep. PMID 32956407
- [Derived] Mah JK, Clemens PR, Guglieri M, Smith EC, Finkel RS, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, McDonald CM, Damsker JM, Schwartz BD, Mengle-Gaw LJ, Jackowski S, Stimpson G, Ridout DA, Ayyar-Gupta V, Baranello G, Manzur AY, Muntoni F, Gordish-Dressman H, Leinonen M, Ward LM, Hoffman EP, Dang UJ; NorthStar UK Network and CINRG DNHS Investigators. Efficacy and Safety of Vamorolone in Duchenne Muscular Dystrophy: A 30-Month Nonrandomized Controlled Open-Label Extension Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2144178. doi: 10.1001/jamanetworkopen.2021.44178. PMID 35076703
- See also: Link to publication — https://pubmed.ncbi.nlm.nih.gov/32956407/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level Group 1: Participants enrolled in Dose Level Group 1 will receive vamorolone 0.25 mg/kg/day.
  Vamorolone 0.25 mg/day/day: Oral administration of 0.25 mg/kg/day daily
- Dose Level Group 2: Participants enrolled in Dose Level Group 2 will receive vamorolone 0.75 mg/kg/day.
  Vamorolone 0.75 mg/day/day: Oral administration of 0.75 mg/kg/day daily
- Dose Level Group 3: Participants enrolled in Dose Level Group 3 will receive vamorolone 2.0 mg/kg/day.
  Vamorolone 2.0 mg/day/day: Oral administration of 2.0 mg/kg/day daily
- Dose Level Group 4: Participants enrolled in Dose Level Group 5 will receive vamorolone 6.0 mg/kg/day.
  Vamorolone 6.0 mg/day/day: Oral administration of 6.0 mg/kg/day daily
Period: Overall Study
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Started | 11 | 12 | 12 | 11
Completed | 10 | 11 | 11 | 9 (Subjects escalated from lower dose groups)
Not Completed | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Subjects entered this study in one of 4 dose level groups, but were allowed to escalate/de-escalate during the course of the study.
Groups:
- Dose Level Group 4: Participants enrolled in Dose Level Group 4 will receive vamorolone 6.0 mg/kg/day.
  Vamorolone 6.0 mg/day/day: Oral administration of 6.0 mg/kg/day daily
- Total: Total of all reporting groups
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4 | Total
Number analyzed (Participants) | 11 | 12 | 12 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.87 (1.135) | 5.11 (0.805) | 5.13 (.964) | 5.27 (0.856) | 5.33 (0.965)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 11 | 12 | 12 | 11 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 11 | 11 | 12 | 8 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 10 | 10 | 12 | 11 | 43
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 2 | 2 | 7
  Sweden | 0 | 4 | 0 | 0 | 4
  United States | 8 | 3 | 2 | 5 | 18
  United Kingdom | 0 | 0 | 4 | 2 | 6
  Israel | 0 | 3 | 2 | 0 | 5
  Australia | 0 | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE Version 4.03
Description: To evaluate the long-term safety and tolerability of vamorolone, administered orally at daily doses up to 6.0 mg/kg/day over a 24- month Treatment Period, in boys ages 4-7 years with DMD; Treatment-emergent adverse events (TEAEs) are defined as any adverse event or worsening of an existing conditions after initiation of the investigational product and through the subject's last study visit (study completion or early termination);
Time Frame: 24 months
Population: All subjects who receive at least one dose of vamorolone study medication in the study will be included in the Safety Population. The Safety Population is the primary analysis population for safety assessments.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level Group 4: Participants enrolled in Dose Level Group 4 will receive vamorolone 4.0 mg/kg/day.
  Vamorolone 4.0 mg/day/day: Oral administration of 4.0 mg/kg/day daily
- Dose Level Group 5: Participants enrolled in Dose Level Group 5 will receive vamorolone 6.0 mg/kg/day.
  Vamorolone 6.0 mg/day/day: Oral administration of 6.0 mg/kg/day daily
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4 | Dose Level Group 5
Number analyzed (Participants) | 11 | 23 | 38 | 3 | 41
Participants | 4 | 14 | 29 | 1 | 39

2. Primary Outcome: Total Number of Adverse Events as Assessed by CTCAE Version 4.03
Description: To evaluate the long-term safety and tolerability of vamorolone, administered orally at daily doses up to 6.0 mg/kg/day over a 24-month Treatment Period, in boys ages 4-7 years with DMD. Treatment-emergent adverse events (TEAEs) are defined as any adverse event or worsening of an existing conditions after initiation of the investigational product and through the subject's last study visit (study completion or early termination).
Time Frame: 24 Months
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4 | Dose Level Group 5
Number analyzed (Participants) | 11 | 23 | 38 | 3 | 41
Events
  Total Number of AEs | 15 | 34 | 203 | 5 | 302
  Total Number of TEAEs | 14 | 34 | 202 | 5 | 300

ADVERSE EVENTS:
Time Frame: Adverse events, including Serious Adverse Events (SAEs), and concomitant medications will be assessed at each study visit and recorded throughout the 24 months treatment period.
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4 | Dose Level Group 5
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/23 | 0/38 | 0/3 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/23 | 0/38 | 0/3 | 1/41
Other Adverse Events (participants affected / at risk) | 4/11 | 14/23 | 29/38 | 1/3 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level Group 1 (N=11) | Dose Level Group 2 (N=23) | Dose Level Group 3 (N=38) | Dose Level Group 4 (N=3) | Dose Level Group 5 (N=41)
Pneumonia (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0
Myoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level Group 1 (N=11) | Dose Level Group 2 (N=23) | Dose Level Group 3 (N=38) | Dose Level Group 4 (N=3) | Dose Level Group 5 (N=41)
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 5 | 0 | 4
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 5 | 1 | 7
Chest Pain (General disorders) | 0 | 1 | 1 | 0 | 3
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 9 | 0 | 8
Ear Infection (Infections and infestations) | 0 | 1 | 2 | 0 | 4
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Influenza (Infections and infestations) | 0 | 1 | 3 | 0 | 6
Nasopharyngitis (Infections and infestations) | 0 | 1 | 7 | 0 | 12
Otitis media (Infections and infestations) | 0 | 0 | 3 | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 2 | 2 | 0 | 3
Upper respiratory tract infection (General disorders) | 0 | 2 | 5 | 0 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 0 | 6
Weight increased (Investigations) | 0 | 0 | 2 | 0 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5 | 0 | 6
Headache (Nervous system disorders) | 0 | 0 | 4 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 7 | 0 | 8
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 3
Lipids Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 2 | 0 | 0
Body Tinea (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Medical device site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Medical device site rash (General disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03038399/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03038399/SAP_002.pdf
  • Informed Consent Form (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03038399/ICF_001.pdf